CLINICAL TRIAL: NCT00672698
Title: Evaluation of Surgical Risk in Elderly Patients Submitted to Elective Surgery: Comparative Study of Elective Vascular, Digestive and Biliary Surgery
Brief Title: Evaluation of Surgical Risk in Elderly Patients Submitted to Elective Surgery
Status: Withdrawn | Type: Observational
Why Stopped: NOT ENOUGH DATA AVAILABLE
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Principal Investigator, MARCELO A. BELTRAN, M.D., DIGESTIVE SURGEON, Cirujanos la Serena
Other Study IDs: 15042008/001
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: PERIPHERAL VASCULAR DISEASES; Digestive Diseases; BILIARY TRACT DISEASES
Keywords: SURGICAL RISK; ELDERLY; MAJOR SURGERY; P-POSSUM; SAPS II
MeSH Terms: conditions — Peripheral Vascular Diseases; Digestive System Diseases; Biliary Tract Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- I: VASCULAR SURGERY
  Interventions: Procedure: SURGERY
- II: DIGESTIVE SURGERY
  Interventions: Procedure: SURGERY
- III: BILIARY TRACT SURGERY
  Interventions: Procedure: SURGERY

INTERVENTIONS:
Procedure: SURGERY — ELECTIVE SURGICAL PROCEDURES

SUMMARY:
The purpose of this study is to establish the surgical risk factors and differences between different diseases in elderly patients submitted to elective surgery in our institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years of age
* All necessary data to calculate p-possum and saps II

Exclusion Criteria:

* Patients with incomplete data

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients older than 65 years of age submitted to elective surgery at our institution
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 YEAR

SECONDARY OUTCOMES:
Morbidity | 1 MONTH

CONTACTS AND LOCATIONS:
Overall Officials: Marceloa A Beltran, M.D., Principal Investigator — Hospital de La Serena
Locations (1):
- Hospital De La Serena, La Serena, Coquimbo Region, Chile